CLINICAL TRIAL: NCT01327313
Title: A Phase I, Open-label Trial to Investigate the Safety, Tolerability, and Pharmacokinetics of EMD525797 After Single Dose and Repeated Dosing at Different Dose Levels in Japanese Patients With Advanced or Metastatic Solid Tumors and Progressive Diseases Following Prior Chemotherapy
Brief Title: A Study of EMD525797 in Solid Tumor Patients in Japan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200017-007
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Solid Tumor
Keywords: alpha v integrin; antibody; solid tumor; Japanese; EMD525797

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- EMD525797 250 milligram (mg) (Experimental)
  Interventions: Biological: EMD525797
- EMD525797 500 mg (Experimental)
  Interventions: Biological: EMD525797
- EMD525797 1000 mg (Experimental)
  Interventions: Biological: EMD525797
- EMD525797 1500 mg (Experimental)
  Interventions: Biological: EMD525797

INTERVENTIONS:
Biological: EMD525797 — Subjects will receive 250 milligram (mg) of EMD525797 intravenously every 2 weeks, until progressive disease (PD), unacceptable toxicity or withdrawal of consent.
  Arms: EMD525797 250 milligram (mg)
Biological: EMD525797 — Subjects will receive 500 mg of EMD525797 intravenously every 2 weeks, until PD or unacceptable toxicity or withdrawal of consent.
  Arms: EMD525797 500 mg
Biological: EMD525797 — Subjects will receive 1000 mg of EMD525797 intravenously every 2 weeks, until PD or unacceptable toxicity or withdrawal of consent.
  Arms: EMD525797 1000 mg
Biological: EMD525797 — Subjects will receive 1500 mg of EMD525797 intravenously every 2 weeks, until PD or unacceptable toxicity, or withdrawal of consent.
  Arms: EMD525797 1500 mg

SUMMARY:
The primary objectives are to assess the safety and tolerability of single and repeated doses of EMD525797, and characterize Pharmacokinetics (PK). The secondary objectives are to investigate the immunogenicity and Progressive disease (PD), and to assess the anti-tumor activity of EMD525797.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to (>=) 20 years
* Histologically or cytologically proven advanced or metastatic solid tumor
* Evidence of progressive disease after standard chemotherapy or no standard chemotherapy
* Confirmation of availability of formalin-fixed paraffin-embedded (FFPE) tumor block(s) or tissue sections
* Presence of at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0 complete tumor assessment to be performed within the 30 days prior to the first EMD525797 administration
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Estimated life expectancy of at least 3 months
* Absolute Neutrophil Count (ANC) >= 1.5 x 10^9 per liter (/Liter)
* Platelets >= 100 x 10^9/Liter
* Haemoglobin >= 9.0 gram per deciliter (g/dL) (without transfusions)
* Total bilirubin less than or equal to (<=) 1.5 x upper limit of normal (ULN)
* Aspartate transaminase (AST), alanine transaminase (ALT) less than or equal to (<=) 3 x ULN
* In subjects with hepatic metastasis, total bilirubin <= 3 x ULN, AST and ALT <= 5 x ULN
* Prothrombin time (PT), prothrombin time/international normalized ratio (PT/INR), and activated partial thromboplastin time (APTT) within normal limits
* Creatinine clearance >= 50 milliliter per minute (mL/min)

Other protocol defined inclusion criteria could also apply

Exclusion Criteria:

* Previous treatment with anti-integrin therapy
* Radiotherapy to bone lesions, systemic surgery, orthopedic surgery (all within the 4 week prior to treatment with EMD525797), clinically significant unhealed wound, or unrecovered bone fracture
* Chronic doses of oral steroids, defined as >= 10 milligram of prednisone equivalents per day
* Confirmed or clinically suspected brain or leptomeningeal metastases
* Known hypersensitivity to EMD525797 or its excipients
* History of allergic reactions to other monoclonal antibody therapy
* Antibody treatment within the past 8 weeks or chemotherapy within the 4 weeks prior to treatment with EMD525797
* Uncontrolled diabetes
* Uncontrolled hypertension defined as systolic blood pressure >= 160 millimeter of mercury (mmHg) and/or diastolic blood pressure >= 100 millimeter of mercury (mmHg) under resting conditions
* Autoimmune diseases
* Current history of chronic daily acetylsalicylic acid (ASS) therapy (ASS at doses <=100 mg is permitted)
* Bleeding disorders;
* History of thromboembolic events (history of superficial thrombophlebitis is not an exclusion
* Anticoagulants within the past 10 days prior to the first treatment and during treatment period
* Severe peripheral vascular disease or ulceration
* Unstable angina pectoris, or myocardial infarction or other severe heart diseases within the past 6 months before treatment with EMD 525797
* Clinical significant abnormal ECG at screening
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Known HIV infection, active or chronic carrier of hepatitis B virus (HBV antigen positive or HBV DNA positive) or hepatitis C virus (HCV antibody positive)

Other protocol defined exclusion criteria could also apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., Japan
Locations (1):
- For Recruiting, Locations in, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- EMD525797 250 mg: 250 milligram (mg) of EMD525797 was administered as an intravenous infusion over 1 hour every 2 Weeks until progressive disease (PD), unacceptable toxicity, or withdrawal of consent.
- EMD525797 500 mg: 500 mg of EMD525797 was administered as an intravenous infusion over 1 hour every 2 Weeks until progressive disease (PD), unacceptable toxicity, or withdrawal of consent.
- EMD525797 1000 mg: 1000 mg of EMD525797 was administered as an intravenous infusion over 1 hour every 2 Weeks until progressive disease (PD), unacceptable toxicity, or withdrawal of consent.
- EMD525797 1500 mg: 1500 mg of EMD525797 was administered as an intravenous infusion over 1 hour every 2 Weeks until progressive disease (PD), unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Started | 8 | 6 | 6 | 7
Completed | 8 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The all-subjects set included all the subjects who signed the informed consent and were treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 7 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (11.64) | 60.5 (4.42) | 54.7 (14.32) | 57.3 (10.81) | 56.3 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 4 | 12
  Male | 6 | 3 | 3 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose-limiting Toxicities (DLTs)
Description: DLT was defined as any Grade 3 or 4 haematological or non-haematological toxicity occurring at any dose level until the end of Week 4, and suspected to be reasonably related to the investigational medicinal product by the Investigator and/or Sponsor. Toxicities not considered to be DLTs are as follows- Allergic reactions or anaphylaxis; any Grade 3 or 4 out-of-range laboratory values without any clinical correlate, which were reversible within 7 days, unless the Investigator decided this event is clinically significant. For this reason Grade 3 or 4 out-of-range laboratory values must be re-assessed within 7 days. In case the Investigator provides the subject any treatment(s) due to the out-of-range laboratory values, the event was regarded as a DLT.
Time Frame: Baseline up to Week 4
Population: Dose escalation analysis set/DLT analysis set included all subjects who experienced a DLT or subjects who did not experience a DLT and had a relative dose intensity of >= 75 percent (%) during the DLT observation period.
Measure: Number; unit: subjects
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6
subjects | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax): After Single Dose
Time Frame: Pre-dose, hour 1(end of infusion [EOI]), 4, 8, 24, 48, and 96 hours after start of infusion at Week 1
Population: The pharmacokinetic (PK) analysis set included all subjects who received at least the first dose of the study drug and who provided sufficient data for a concentration-time profile for EMD 525797.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
microgram per milliliter (mcg/mL) | 73.12 (12.1) | 162.48 (15.2) | 419.26 (16.4) | 683.46 (28.0)

3. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of EMD 525797:After Multiple Dose
Time Frame: Pre-dose, hour 1 (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: The PK analysis set included all subjects who received at least the first dose of the study drug and who provided sufficient data for a concentration-time profile for EMD 525797. Here N (number of subjects analyzed) signifies the total number of subjects evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL | 89.336 (6.6) | 198.728 (20.1) | 680.022 (18.1) | 1170.73 (22.2)

4. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration(AUC0-t) of EMD 525797: After Single Dose
Description: Area under the serum concentration-time curve from time zero to the last sampling time at which the concentration is at or above Lower limit of quantification (LLQ).
Time Frame: Pre-dose, hour 1 (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 1
Population: The PK analysis set included all subjects who received at least the first dose of the study drug and who provided sufficient data for a concentration-time profile for EMD 525797.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*mcg/mL
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
hour*mcg/mL | 7942.6 (19.6) | 21562.3 (14.0) | 67545.6 (18.9) | 95369.6 (40.9)

5. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration(AUC0-t) of EMD 525797: After Multiple Dose
Description: Area under the serum concentration-time curve from time zero to the last sampling time at which the concentration is at or above LLQ.
Time Frame: Pre-dose, hour 1 (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*mcg/mL
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour*mcg/mL | 10674.2 (30.2) | 37344.9 (28.2) | 159979.5 (29.5) | 242989.3 (35.7)

6. Primary Outcome: Total Body Clearance (CL) of EMD 525797: After Single Dose
Description: Total body clearance of drug in serum was calculated: as CL= Dose divided by Area under the serum concentration-time curve from time zero to infinity (AUC0-inf).
Time Frame: Pre-dose, hour 1 (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
liter per hour | 0.0294 (24.5) | 0.0188 (29.9) | 0.0083 (23.0) | 0.0089 (52.9)

7. Secondary Outcome: Number of Subjects With Overall Tumor Response
Description: Overall tumor response was defined as the presence of at least one confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0. Complete response was defined as the disappearance of all target and non-target lesions and normalization of serum levels of tumor markers. PR is at least a 30 percent (%) decrease in the sum of the longest diameter (LD) of target lesions, taking as a reference the baseline sum LD.
Time Frame: Baseline up to Week 36
Population: Full analysis set included all subjects who received at least one (non-zero) administration of the trial medication.
Measure: Number; unit: subjects
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
subjects | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Subjects With Clinical Benefit
Description: Clinical benefit was defined as presence of at least one confirmed CR, PR, or stable disease (SD) lasting at least 12 weeks according to RECIST v1.0. Per RECIST v1.0: CR was defined as disappearance of all target and non-target lesions and normalization of serum levels of tumor markers . PR was defined as >=30% decrease in sum of longest diameters of target lesions taking as reference baseline sum longest diameters associated to non-progressive disease response for non-target lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference smallest sum of longest dimensions since treatment started associated to non-progressive disease response for non-target lesions.
Time Frame: Baseline up to Week 36
Population: Full analysis set included all subjects who received at least one (non-zero) administration of the trial medication.
Measure: Number; unit: subjects
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
subjects | 0 | 0 | 0 | 0

9. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS time was defined as the time (in months) from the first dosing date to the date of first documentation of disease progression as reported and documented by the Investigator (i.e. radiological progression per RECIST version 1.0) or death for any cause within 12 weeks after last tumor assessment. Subjects without event are censored on the date of last tumor assessment.
Time Frame: From first dosing date until disease progression or death, maximum up to Week 36
Population: Full analysis set included all subjects who received at least one (non-zero) administration of the trial medication.
Measure: Median (Full Range); unit: months
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
months | 1.18 [0.8 to 1.2] | 1.23 [1.2 to 2.1] | 1.31 [1.2 to 5.5] | 1.25 [0.4 to 2.8]

10. Secondary Outcome: Apparent Terminal Half Life (t1/2): After Single Dose
Time Frame: Pre-dose, end of infusion (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 1
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
hour | 83.95 [52.7 to 124.1] | 114.45 [45.6 to 272.4] | 298.99 [205.7 to 411.7] | 240.76 [150.5 to 612.3]

11. Secondary Outcome: Apparent Terminal Half Life (t1/2): After Multiple Dose
Time Frame: Pre-dose, EOI, 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour | 119.58 [56.2 to 145.9] | 195.75 [86.9 to 221.7] | 345.92 [294.0 to 751.1] | 448.45 [224.3 to 760.5]

12. Secondary Outcome: Time to Maximum Observed Serum Concentration (Tmax): After Single Dose
Time Frame: Pre-dose, end of infusion (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 1
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
hour | 1.033 [1.02 to 24.03] | 1.033 [1.00 to 4.00] | 3.967 [1.02 to 7.95] | 1.067 [1.03 to 24.05]

13. Secondary Outcome: Time to Maximum Observed Serum Concentration (Tmax): After Multiple Dose
Time Frame: Pre-dose, EOI, 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour | 1.042 [1.00 to 47.97] | 3.00 [1.02 to 24.12] | 1.025 [1.00 to 4.02] | 4.000 [1.07 to 23.95]

14. Secondary Outcome: Elimination Rate Constant (λz): After Single Dose
Description: The elimination rate constant obtained from linear regression of the terminal phase of the log transformed concentration-time data.
Time Frame: Pre-dose, end of infusion (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
per hour | 0.00895 (31.5) | 0.00573 (66.7) | 0.00237 (25.6) | 0.00272 (49.6)

15. Secondary Outcome: Elimination Rate Constant ( λ z): After Multiple Dose
Description: as for outcome 14
Time Frame: Pre-dose, EOI, 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
per hour | 0.00639 (35.5) | 0.00407 (36.7) | 0.00178 (35.2) | 0.00170 (53.3)

16. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) After Multiple Doses
Description: The observed minimum serum concentration determined directly from the serum concentration-time profile of each subject.
Time Frame: Pre-dose, EOI, 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL | 5.64 (154.6) | 44.22 (40.2) | 200.5 (30.3) | 286.11 (30.5)

17. Secondary Outcome: Observed Serum Concentration Immediately Before Next Dosing (Cpre)
Description: The observed serum concentration immediately before next dosing determined directly from the serum concentration-time profile of each subject (= trough concentration)
Time Frame: Pre-dose, EOI, 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL | 5.73 (150.7) | 44.28 (40.1) | 200.05 (30.3) | 286.11 (30.5)

18. Secondary Outcome: Average Serum Concentration at Steady State (Cav)
Description: The Cav was calculated by dividing the area under the serum concentration-time curve within one complete dosing interval (AUCtau) by the dosing interval (2 weeks or 336 hoursi.e. Cav =AUCtau/tau).
Time Frame: Pre-dose, EOI, 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL | 33.23 (26.4) | 96.91 (26.9) | 395.47 (19.1) | 574.09 (25.1)

19. Secondary Outcome: Area Under the Serum Concentration-time Curve Within One Complete Dosing Interval( AUCtau): After Single Dose
Time Frame: Pre-dose, end of infusion (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*mcg/mL
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
hour*mcg/mL | 7970.1 (20.3) | 21563.6 (14.0) | 67555.4 (19.0) | 100861.0 (26.5)

20. Secondary Outcome: Area Under the Serum Concentration-time Curve Within One Complete Dosing Interval( AUCtau): After Multiple Dose
Time Frame: Pre-dose, EOI, 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*mcg/mL
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour*mcg/mL | 11164.0 (26.4) | 32561.0 (26.9) | 132877.8 (19.1) | 192894.5 (25.1)

21. Primary Outcome: Total Body Clearance at Steady State (CLss) of EMD 525797
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. CL of drug in serum was calculated as : CL= Dose/ AUC0-inf. Area under the serum concentration-time curve from time zero to infinity (AUC0-inf), calculated as AUC0-t + AUCextra. AUCextra represents an extrapolated value obtained by Clast / λz, where Clast is the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above LLQ and λz is the elimination rate constant.
Time Frame: Pre-dose, hour 1 (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
liter per hour | 0.0224 (26.4) | 0.0154 (26.9) | 0.0075 (19.1) | 0.0078 (25.1)

22. Primary Outcome: Apparent Volume of Distribution (Vz): After Single Dose
Description: Apparent volume of distribution during the terminal phase, calculated as Vz = Dose/AUC0-inf multiplied by elimination rate constant [λz]) following single dose. Area under the serum concentration-time curve from time zero to infinity, calculated (AUC0-inf) as AUC0-t + AUCextra. AUCextra represents an extrapolated value obtained by Clast / λz, where Clast is the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above LLQ and λz is the elimination rate constant. And the elimination rate constant obtained from linear regression of the terminal phase of the log transformed concentration-time data. A minimum of three points is required to calculate λz.
Time Frame: Pre-dose, hour 1 (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
liter | 3.285 (20.5) | 3.284 (37.8) | 3.506 (23.7) | 3.268 (17.3)

23. Primary Outcome: Pharmacokinetics of EMD 525797 - Trough Values
Description: as for outcome 17
Time Frame: Pre-dose, hour 1 (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL | 5.73 (150.7) | 44.28 (40.1) | 200.05 (30.3) | 286.11 (30.5)

24. Primary Outcome: Apparent Volume of Distribution: After Multiple Dose
Description: Apparent volume of distribution during the terminal phase, calculated as Vz = Dose/(Area under the serum concentration-time curve within one complete dosing interval [AUCtau]* λz) following multiple dose.
Time Frame: Pre-dose, hour 1 (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
liter | 3.505 (18.2) | 3.775 (22.0) | 4.224 (21.5) | 4.565 (40.0)

25. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) was the apparent volume of distribution at steady-state.
Time Frame: Pre-dose, EOI, 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
liter | 3.584 (9.6) | 4.004 (17.2) | 4.131 (21.6) | 4.392 (38.9)

26. Secondary Outcome: Mean Residency Time (MRT0-inf)
Description: MRT0-inf of drug in the body was calculated by dividing the area under the first moment curve from time zero to infinity with area under the first moment curve from time zero to infinity minus half of infusion of duration (MRT0-inf = AUMC0-inf/AUMC0-inf - T/2).
Time Frame: Pre-dose, end of infusion (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 7
hour | 118.46 (25.0) | 187.29 (48.7) | 408.34 (23.3) | 357.21 (48.8)

27. Secondary Outcome: Mean Residence Time at Steady State (MRTss)
Description: MRTss = (AUMCtau + tau(AUCinf - AUCtau))/ AUCtau) - T/2, where AUMCtau was the area under the first moment curve within one complete dosing interval and T was the infusion duration. Area under the serum concentration-time curve from time zero to infinity, calculated as AUC0-t + AUCextra. AUCextra represents an extrapolated value obtained by Clast / λz, where Clast is the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above LLQ and λz is the elimination rate constant.
Time Frame: Pre-dose, EOI, 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour | 160.05 (28.0) | 260.73 (29.5) | 548.88 (35.5) | 564.86 (53.1)

28. Secondary Outcome: Percentage Peak-Trough Fluctuation (PTF)
Description: The peak trough fluctuation over one dosing interval at steady state, calculated as PTF (%) = ( [Cmax - Cmin] / Cav ) multiplied by 100.
Time Frame: Pre-dose, EOI, 4, 8, 24, 48, and 96 hours after start of infusion at Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage fluctuation
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage fluctuation | 243.64 (33.4) | 157.93 (17.0) | 118.69 (31.8) | 153.22 (20.7)

29. Secondary Outcome: Accumulation Ratio (Rac)
Description: Accumulation ratio for AUC, calculated as area under the serum concentration-time curve within one complete dosing interval at 3rd infusion divided by area under the serum concentration-time curve within one complete dosing interval at 1st infusion.
Time Frame: Pre-dose, end of infusion (EOI), 4, 8, 24, 48, and 96 hours after start of infusion at Week 1 and Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ratio | 1.371 (23.5) | 1.510 (18.4) | 1.967 (13.0) | 1.762 (12.0)

ADVERSE EVENTS:
Time Frame: First dose of the study drug up to 31+/-3 days after the last administration of EMD 525797, assessed upto maximum of 22 months.
Description: The safety analysis set included all subjects who received at least one (non-zero) administration of the trial medication.
Arm/Group | EMD525797 250 mg | EMD525797 500 mg | EMD525797 1000 mg | EMD525797 1500 mg
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/6 | 1/6 | 1/7
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMD525797 250 mg (N=8) | EMD525797 500 mg (N=6) | EMD525797 1000 mg (N=6) | EMD525797 1500 mg (N=7)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMD525797 250 mg (N=8) | EMD525797 500 mg (N=6) | EMD525797 1000 mg (N=6) | EMD525797 1500 mg (N=7)
Anaemia Of Malignant Disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 3 (4) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (6)
Pyrexia (General disorders) | 3 (5) | 1 (1) | 1 (1) | 1 (2)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Calcium Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Mb Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophil Count Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibrin D Dimer Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No